CLINICAL TRIAL: NCT04121364
Title: Immediate Placement and Stabilization of Dental Implants With Tetranite® Stabilization Material in Mandibular and Maxillary Tooth Extraction Sites That Fail to Provide Adequate Primary Stability
Brief Title: Immediate Placement and Stabilization of Dental Implants With Tetranite Stabilization Material in Mandibular and Maxillary Tooth Extraction Sites That Fail to Provide Adequate Primary Stability
Status: Completed | Type: Interventional
Sponsor: RevBio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DVAL18041
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Results first posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-08

CONDITIONS: Adhesive Dental

STUDY DESIGN:
Intervention Model Description: Non randomized, single arm, objective performance criteria study
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Tetranite (Experimental): All patients enrolled in study will receive the dental adhesive with a dental implant. The robustness of the dental implant stability will be assessed at various time points.
  Interventions: Device: Tetranite

INTERVENTIONS:
Device: Tetranite — Dental Adhesive for increased implant stability

SUMMARY:
This study is to determine if a new bone adhesive is useful in stabilizing dental tooth implants. Data collected from the study will examine the strength, performance, and the safety of the material.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single arm, pilot clinical study evaluating the use of TN-SM for implant stabilization immediately after tooth extraction. The purpose of this pilot study is to test performance characteristics and capabilities of study design, recruitment criteria, procedures, measures, and operational strategies that are under consideration for use in a subsequent, larger clinical pivotal study. The purpose of the subsequent study will be to provide data demonstrating the safety and efficacy for the use of TN-SM to provide immediate and continued stabilization of implants placed into otherwise unstable sites. Use of TN-SM eliminates the need for the standard practice of bone grafting after tooth extraction and staged implant placement, significantly shortening the overall length of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent;
* 21+ Age;
* Require tooth extraction and replacement with dental implant;
* Have opposing dentition;
* Committed to Study and Follow-up period;
* ASA I or II;
* Planned "implant site" must have 1 adjacent tooth;
* Sufficient bone Height for safe dental implant placement;
* At least 2 mm of apical bone for seating of implant.

Exclusion Criteria:

* Any significant disease that would preclude a dental implant
* Any oral surgery contraindications
* Subjects with mucosal Disease
* Subjects with bone diseases or conditions (e.g. Paget's disease, fibrous dysplasia, history of osteomyelitis, etc.) in the region of the potential study implant site;
* Subjects with a history of local radiation therapy in the head/neck area or osteonecrosis of the jaws;
* Subjects with any acute and untreated endodontic lesions or periodontal disease;
* Subjects receiving, or having a recent or long-term history of receiving, oral or parenteral anti-osteoclastic agents [e.g., bisphosphonates, Xgeva® and Prolia® (denosumab); Forteo® (teriparatide), strontium ranelate, etc.], or anti-angiogenesis factors;
* Subjects who have major active substance abuse problems (e.g., alcoholism, opiate addiction, methamphetamine abuse, etc.);
* Subjects who are pregnant or intending to become pregnant during the duration of the study;
* Subjects who are heavy smokers (defined as >10 cigarettes per day or >1 cigar per day or equivalent of electronic cigarette vaping) or chew tobacco;
* Subjects with inadequate oral hygiene or who are unmotivated for adequate home care;
* Subjects who have physical or mental handicaps that would interfere with the ability to perform adequate oral hygiene;
* Subjects who have undergone administration of any investigational device within 30 days of enrollment in the study;
* Subjects who are allergic or otherwise sensitive to any materials likely encountered during the course of the study (e.g. titanium, suture materials, local anesthetics);
* Subjects with conditions or circumstances, which, in the opinion of the Investigator, would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance or unreliability
* Any site into which the implant is not or cannot be placed during the same visit as the extraction;
* Any implant site where there is a dehiscence or fenestration of buccal or lingual plates of bone greater than 5mm in any direction.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2023-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center - San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tetranite
Started | 20
Completed | 6
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Tetranite
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.05 (13.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Implant Success (Modified Buser Criteria)
Description: The primary endpoint is a composite measure of implant success (after criteria of Buser, et. al.1) at six-month post-functional loading consisting of:
  * Presence of the implant at its site of implantation; and,
  * Absence of a recurrent peri-implant infection with suppuration; and,
  * Absence of mobility, defined as:
    * Lack of implant rotation subjected to 20 Ncm of clockwise torque applied 15 minutes after implant placement; and.
    * Lack of implant rotation subjected to 35 Ncm of clockwise torque applied 13 weeks after implant placement; and,
    * No construct mobility upon palpation at 6 months post-functional loading; and,
  * Absence of encapsulation defined as continuous radiolucency around the implant in a periapical radiograph.
Time Frame: 6 months
Population: Surviving implants assessed. Number of subjects meeting the criteria reported
Measure: Number; unit: participants
Arm/Group | Tetranite
Number analyzed (Participants) | 9
participants | 6

2. Secondary Outcome: Adverse Events (Serious, Device Related)
Description: Incidence of Device related Serious adverse events
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study: from device/implant placement through the 24 month post-loading follow-up. Additionally, patients who experienced an implant failure were followed for adverse events through 12 months post-implant failure.
Arm/Group | Tetranite
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 13/20
Other Adverse Events (participants affected / at risk) | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tetranite (N=20)
Implant Loss (Infections and infestations) | 13 (13) — Implant loss following mobility, infection, and/or bone loss.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tetranite (N=20)
Suppuration (Infections and infestations) | 4 (10) — Suppuration near/around the implant site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT04121364/Prot_SAP_000.pdf